CLINICAL TRIAL: NCT06776003
Title: Continuous Mobility and Physical Activity in Vertebroplasty vs Sham for Osteoporotic Vertebral Fracture: a Single-center, Double-blind Randomized Controlled Clinical Trial
Brief Title: Continuous Mobility and Physical Activity in Vertebroplasty vs Sham for Osteoporotic Vertebral Fracture
Acronym: VOPE2 COMPAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23/40938; 112199 (Registry Identifier: Den Videnskabsetiske Komité for Region Syddanmark)
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Osteoporotic Vertebral Compression Fractures
Keywords: Accelerometer; Global Positioning System; Vertebroplasty; Physical Activity; Mobility; Osteoporosis; Spinal Surgery; ActiGraph; Accelerometry; GPS; Osteoporotic
MeSH Terms: conditions — Motor Activity; Osteoporosis | interventions — Vertebroplasty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vertebroplasty (Active Comparator): Polymethyl-methacrylate (PMMA) cement is prepared and injected slowly into the vertebral body under constant bi-plane fluoroscopy
  Interventions:
  Procedure: Vertebroplasty
  Interventions: Procedure: Vertebroplasty
- Sham vertebroplasty (Sham Comparator): A short needle is passed through the skin, but not as far as the periosteum. PMMA is mixed to mimic the PVP procedure but not injected into the vertebral body.
  Interventions:
  Procedure: Sham Vertebroplasty
  Interventions: Procedure: Sham Vertebroplasty

INTERVENTIONS:
Procedure: Vertebroplasty — Polymethyl-methacrylate (PMMA) cement is injected slowly into the vertebral body under constant bi-plane fluoroscopy
  Other Names: Percutaneous vertebroplasty; PVP
  Arms: Vertebroplasty
Procedure: Sham Vertebroplasty — A short needle is passed through the skin, but not as far as the periosteum. PMMA is mixed to mimic the PVP procedure but not injected into the vertebral body.
  Arms: Sham vertebroplasty

SUMMARY:
The aim of this clinical trial is to determine if vertebroplasty is an effective treatment for acute, painful vertebral fractures due to osteoporosis.

The focus of the study is on the physical activity and mobility of participants.

The main questions the trial aims to answer are:

* Does vertebroplasty lead to increased physical activity as measured by accelerometer?
* Does vertebroplasty lead to increased mobility as measured by GPS (global positioning system)?
* Do physical activity and mobility correlate with pain, disability and quality of life?

Researchers will compare vertebroplasty to sham (simulated surgery without active intervention) to understand if vertebroplasty improves physical activity and mobility.

Participants will

* Undergo vertebroplasty or sham procedure
* Wear an accelerometer and a GPS-reciever in a belt for 1 week before to 4 weeks after the surgery
* Answer questionnaires regarding pain, disability and quality of life at regular intervals.

The knowledge gained from this can help determine who would benefit from vertebroplasty.

DETAILED DESCRIPTION:
Despite attempts at prevention, osteoporotic vertebral fracture occurs with increasing frequency as lifespans increase.

Patients with this disease can experience severe pain and disability, and when conservative treatment is inadequate, vertebroplasty is an option.

In this surgical procedure, polymethyl metacrylate, or "bone cement" is injected into the fractured vertebral body. However, the procedure is currently controversial for the treatment of osteoporotic vertebral fractures because there is not yet consensus on the efficacy.

By investigating the effect of vertebroplasty on mobility and physical activity, this study aims to contribute to resolution of the controversy.

The study is a prospective, double-blind, randomized, sham-controlled clinical trial, where participants will be randomized to either vertebroplasty or a sham operation.

The study is embedded in the ongoing trial "Percutaneous Vertebroplasty Vs. Sham for Osteoporotic Vertebral Compression Fractures Focusing on Pain and Economy (VOPE2)" with ClinicalTrials.gov ID NCT06141187.

A subset of the participants in VOPE2 will, in addition to previously planned activities, be equipped with wearable accelerometers and a global positioning system (GPS).

The trial is designed in accordance with the SPIRIT guidelines.

Potential participants will be identified by referral to the Center for Spine Surgery and Research from general practitioners, chiropractor, physiotherapist, or from hospital inpatient and emergency departments in the region of Southern Denmark.

Participants will then be examined in an outpatient clinic by a spine surgeon, and have MRI scans and X-ray images analyzed by experienced neuro-radiologists.

If eligible, they will be offered to participate following informed consent. An accelerometer and GPS-reciever attached to an elastic waist band are initiated following inclusion.

Subjects will initially be stratified into two groups based on the number of OVCFs into 1-2 levels or 3-4 levels.

Within each of these two groups, randomization sheets in varying blocks of 8 with an equal number of PVP and sham patients in each block will be generated using software (www.randomizer.org) and will be placed in numbered, opaque, sealed envelopes.

Treatment group assignment is 1:1 and will be performed by a scrub nurse in the surgical theatre after the patient is draped but prior to skin incision.

Throughout the trial, only the surgeon and the OR-nurse will have knowledge of the treatment assignment.

The patient and all assessors remain blinded to the treatment group throughout the study. Spine surgeons who are experienced in PVP will perform the surgical procedures.

Anaesthesiologists and spine surgeons are present at the facility in case of complications, following recommendations by the National Health Authority and have the capacity/capability to decompress the spinal canal in case of cement leakage

Based on qualitative studies and clinical experience, patients with painful osteoporotic vertebral fractures restrict their movement because of pain.

This in turn leads to reduced physical activity and diminished ability to move oneself around and away from home, defined here as mobility.

If vertebroplasty is effective, it is expected to lead to increased physical activity and mobility compared to sham, and the outcomes derived from accelerometers and GPS-recievers can supplement patient reports due to their continuous and objective nature.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50+ and diagnosed with symptomatic osteoporotic spinal compression fractures between T6 and L5 (incl).
* Focal tenderness on the level of the vertebral fracture.
* Fractures verified with oedema of the relevant vertebra on the MRI STIR sequence.
* Osteoporotic Fractures type 1-4.
* Fracture involves no more than 4 vertebral body levels.
* Vertebroplasty can be done in one session.
* Back pain score measured on a Visual Analog Scale (VAS, 0 to 100) ≥ 60.
* Able to understand and read Danish.
* Written informed consent.
* Relevant pain started ≤ 3 months prior to enrollment.

Exclusion Criteria:

* Contra-indications for spine surgery.
* Platelets < 30 mia/l.
* Osteoporotic Fractures type 5 and Pincer-type.
* Complete collapse of the vertebral body precluding insertion of needle.
* Presence of neurologic deficit.
* Contraindications for MRI scanning.
* Psychological or psychiatric disorder that is expected to interfere with compliance.
* Active malignancy.
* Mini Mental State Examination (MMSE) test score below 24.
* History of chronic back pain requiring ongoing opiate use.
* Systemic or local infection of the spine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity before and after intervention | One week preoperatively to the end of the fourth postoperative week.
  Physical activity is measured by accelerometer and presented as mean ENMO (euclidian norm minus one) and mean TAC/d (total activity count per day).
  An unweighted average of valid days within the preoperative week is compared with the unweighted average of valid days within the four postoperative weeks by relative change in percent.

SECONDARY OUTCOMES:
Daily and weekly physical activity | One week preoperatively to 4 weeks postoperatively
  Physical activity is measured by accelerometer and presented as difference in mean ENMO (euclidian norm minus one) and mean TAC/d (total activity count per day). Daily means are based on valid wear-time. Weekly means are calculated as unweighted averages of all valid days within the week.
Change in daily and weekly physical activity | One week preoperatively to 4 weeks postoperatively
  Physical activity is measured by accelerometer and presented as difference in mean ENMO (euclidian norm minus one) and mean TAC/d (total activity count per day). Daily means are based on valid wear-time. Weekly means are calculated as unweighted averages of all valid days within the week.
  This outcome supplements the primary outcome to cover changes within the full study period. Changes are reported as relative percentages.
Physical activity levels | One week preoperatively to 4 weeks postoperatively
  Based on cut-points applied to the ENMO or count measurements, the valid wear-time is divided into intensity classes "sedentary", "light activity" or "moderate to vigorous activity". Time spent in each class is presented as percentage of valid wear-time.
Change in physical activity levels | One week preoperatively to 4 weeks postoperatively
  Based on cut-points applied to the ENMO or count measurements, the valid wear-time is divided into intensity classes "sedentary", "light activity" or "moderate to vigorous activity". Time spent in each class is presented as percentage of valid wear-time and changes as absolute percentage points.
Total daily distance and change in total daily distance | One week preoperatively to 4 weeks postoperatively
  Total daily distance traveled in meters based on GPS positions. Changes are relative in percentages.
Time spent stationary and change in time spent stationary | One week preoperatively to 4 weeks postoperatively
  Percentage of time spent stationary based on GPS positions relative to the days' recording. Change is absolute percentage points.
Time spent away from home and change in time spent away from home | One week preoperatively to 4 weeks postoperatively
  Percentage of time per day where the GPS records a position away from home relative to the days' recordings. Change is in absolute percentage points.
Patient-reported pain intensity. | VAS will be recorded once preoperatively and again 1, 2, 3, 4 and 5 days + 2 and 4 weeks postoperatively.
  Pain intensity over the previous 24 hours using the 100-point visual analog scale, where 0 is no pain and 100 is the worst imaginable pain.
Patient-reported disability | Preoperatively and at 4 weeks postoperatively
  The patients rate their disability using the Oswestry Disability Index (ODI) questionnaire.
Patient-reported health-related quality of life. | Preoperatively and at 4 weeks postoperatively
  Health-related quality of life. on the EuroQol 5-dimension 5-level (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Ø Andersen, Prof, MD, Study Chair — Spine Centre of Southern Denmark
Locations (1):
- Spine Centre of Southern Denmark, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data from questionnaires, accelerometers and GPS-records will be made available in an anonymized form to researchers who present a proposal for the use that is reasonable and can be approved by the study authors.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The IPD and data will be stored for five years from the completetion of the study at the trial site followed by archiving at the Danish National Archives.
Access Criteria: Researchers can request access to the information by contacting the investigator via email at soren.wittorff.sorensen@rsyd.dk